CLINICAL TRIAL: NCT07366567
Title: Effect of Foot Bath on Pain, Sleep, and Comfort Levels After Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Effect of Foot Bath on Pain, Sleep, and Comfort Levels After Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Zeynep Kızılcık Ozkan, Associate professor, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/284
Record Dates: First submitted 2025-11-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pain, Postoperative; Sleep
Keywords: pain; foot bath; sleep quality; comfort
MeSH Terms: conditions — Pain, Postoperative; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group will receive a foot bath. Patients in the control group will not be intervened within the scope of the study.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (with Foot Bath Device Foot Bath Application (20 min, 41-42°C) (Experimental): Postoperative Preparation: The intervention will commence once the effects of anesthesia have subsided and initial mobilization (routinely 6-8 hours post-surgery) has been achieved. At approximately 9:00 PM, the patient's feet will be prepared by removing socks or adjusting anti-embolic stockings above the ankle . A visual and physical examination of the feet will be conducted to screen for contraindications such as pressure injuries, wounds, or discoloration.
  Foot Bath Intervention: The foot bath procedure will be performed using a disinfected device lined with single-use, watertight bags to ensure hygiene.The water temperature will be strictly maintained at 41-42°C, verified by a non-contact infrared digital thermometer. Both feet will be immersed in the device for a duration of 20 minutes. Post-intervention, the researcher will thoroughly dry the patient's feet and replace their socks or anti-embolic stockings. Any adverse events or side effects observed, recorded.
  Interventions: Other: Foot bath device
- Control group Control group (Standard care (no foot bath procedure) (No Intervention): Patients in the control group will receive routine care. Patient Recruitment and Preoperative Phase: Patients admitted to the General Surgery department for abdominal surgery will be informed about the study on the morning of their procedure. Following the acquisition of both verbal and written informed consent, the Patient Information Form will be completed. To establish a baseline for sleep quality, the Richards-Campbell Sleep Questionnaire (RCSQ) will be administered preoperatively.
  No foot bath application will be in question for the patients in the control group.
  Data Collection and Conclusion: On the morning of the first postoperative day, the RCSQ, GKO (Visual Analog Scale/Global Quality Scale), and pain scores will be administered to evaluate the intervention's impact. The data collection process will conclude following these assessments.

INTERVENTIONS:
Other: Foot bath device — On the day of surgery, patients will receive a foot bath between 9:00 PM and 10:00 PM. Any socks or clothing on both feet will be removed. The feet will be visually and manually examined to determine if they show any signs of illness (pressure ulcers, discoloration, wounds, etc.). The patient will be informed that the foot bath device is disinfected before each use and that water-tight bags will be placed around the device to prevent contact between the foot and the water to facilitate repeated use. The water temperature will be adjusted to 41-42°C using an infrared thermometer (non-contact digital thermometer). Both feet will be placed inside the foot bath device. The patient's feet will remain in the foot bath device for 20 minutes. After the foot bath, the patient's feet will be thoroughly dried with a towel, and the patient will be re-dressed in their existing socks or anti-embolic stockings. Any side effects/adverse reactions, etc., related to the foot bath will be questioned and
  Arms: Experimental group (with Foot Bath Device Foot Bath Application (20 min, 41-42°C)

SUMMARY:
The aim of this study was to investigate the effects of foot bath application on pain level, comfort and sleep quality in the postoperative period.

H1: Foot baths have a postoperative pain-reducing effect. H2: Foot baths have a postoperative comfort-enhancing effect. H3: Foot baths have a postoperative sleep-improving effect.

DETAILED DESCRIPTION:
The research will be conducted with the participation of surgical patients who underwent abdominal surgery between December 2025 and December 2026 in the General Surgery Department of Tekirdag University Hospital.

Using the G*Power 3.1.9.4 program, the minimum number of people to be included in the sample was found to be 88 (44:44), assuming an effect size of 0.8 at a 95% confidence level and a 95% power ratio. To avoid the risk of sample loss, it was decided to include 48 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* who are hospitalized in the General Surgery Clinic,
* are on day 0 of surgery,
* volunteer to participate in the study,
* have no neuropsychiatric diagnosis and are not taking antipsychotic medications,
* are over 18 years of age,
* accept random selection,
* and undergo abdominal surgery.
* For the experimental group, all patients with no infectious diseases (shingles, fungal infections, eczema, warts, calluses), local infections (abscesses, etc.), open lesions/wounds, scar tissue, edema, hematomas, thrombophlebitis, deep vein thrombosis, lymphangitis, coagulation disorders, varicose veins, osteoporosis, osteomyelitis, hepatitis, degenerative joint diseases, neuropathy due to diabetes, toe deformities, recent fractures, dislocations, or ruptures of muscle fibers, tendons, or ligaments will be included in the sample.

Exclusion Criteria:

* patients who underwent multiple simultaneous surgeries along with abdominal surgery,
* those with postoperative complications such as delirium,
* those who underwent reoperation,
* those with a pain score >7 because it could affect sleep levels,
* and those who received narcotic analgesics on postoperative day 0 due to pain will be excluded from the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain level | postoperative period (first day)
  "Numerical rating scale" A score of 0 (zero) indicates no pain, while a score of 10 (ten) indicates unbearable pain.
sleep quality | postoperative period (1st day)
  "The Richards-Campbell Sleep Questionnaire" Each item is scored on a visual analog scale from 0 to 100. Scores between 0 and 25 indicate very poor sleep, while scores between 76 and 100 indicate very good sleep.

SECONDARY OUTCOMES:
Adverse effect | during application and 12 hours of application.
  Adverse effect (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP KIZILCIK ÖZKAN, Assoc.Prof, Study Chair — Trakya University; Ayşe Nur Aktaş, Reg.Nurse, Principal Investigator — Trakya University
Locations (1):
- Trakya University Hospital, Edirne, Cahit Arf Boulevard, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
While obtaining ethics committee approval, the application form included information that the data would only be used by researchers and would not be shared with third parties.

DOCUMENTS (3):
  • Study Protocol (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT07366567/Prot_000.pdf
  • Statistical Analysis Plan (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT07366567/SAP_001.pdf
  • Informed Consent Form (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT07366567/ICF_002.pdf